CLINICAL TRIAL: NCT04598282
Title: A Pilot Study Evaluating Adjunctive Cryopreserved Amniotic Membrane Treatment for Primary or Recurrent Herpes Simplex Dendritic Keratitis
Brief Title: Evaluating Adjunctive Cryopreserved Amniotic Membrane Treatment in Herpes Simplex Dendritic Keratitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patient enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: BioTissue Holdings, Inc (Industry)
Responsible Party: Principal Investigator, Richard Stutzman, MD, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00021203
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Herpes Simplex Dendritic Keratitis
Keywords: Prokera; Adjunctive Cryopreserved Amniotic Membrane; Prokera Slim
MeSH Terms: conditions — Keratitis, Dendritic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (Placebo Comparator): All subjects enrolled in the study will receive the standard of care that includes epithelial debridement of all dendrites via Weck-Cel Cellulose sponge, topical prophylactic antibiotics (e.g., Ocuflox QID (four times daily) for one week) and oral acyclovir (400 mg 5x/day for 10 days for primary cases but tapered to 2x/day for 3 months for recurrent cases based on investigator's discretion).
  Interventions: Other: Standard of Care
- Treatment Arm (Active Comparator): All subjects enrolled in the study will receive the standard of care that includes epithelial debridement of all dendrites via Weck-Cel Cellulose sponge, topical prophylactic antibiotics (e.g., Ocuflox QID for one week) and oral acyclovir (400 mg 5x/day for 10 days for primary cases but tapered to 2x/day for 3 months for recurrent cases based on investigator's discretion). The treatment arm will also receive the placement of PROKERA SLIM for 5-7 days. A second PROKERA SLIM may be applied based on investigator's discretion. For patients with bilateral involvement only the worse eye will be enrolled for the treatment arm.
  Interventions: Device: Prokera Slim

INTERVENTIONS:
Device: Prokera Slim — Placement of an Adjunctive Cryopreserved Amniotic Membrane Treatment.
  Arms: Treatment Arm
Other: Standard of Care — Standard of care includes epithelial debridement of all dendrites via Weck-Cel Cellulose sponge, topical prophylactic antibiotics (e.g., Ocuflox QID for one week) and oral acyclovir (400 mg 5x/day for 10 days for primary cases but tapered to 2x/day for 3 months for recurrent cases based on investigator's discretion).
  Arms: Control Arm

SUMMARY:
To prospectively evaluate the effectiveness of Prokera Slim in adults with primary or recurrent herpetic epithelial keratitis in terms of visual function, corneal opacity, time to resolution, cost of care, number of patient visits.

DETAILED DESCRIPTION:
Cryopreserved amniotic membrane (AM) contains anti-inflammatory, anti-scarring and antiangiogenic effects known in treating many ocular surface diseases. This notion is further strengthened by many studies showing that amniotic membrane can effectively control inflammation in HSV stromal keratitis in a murine model of HSV necrotizing keratitis and surgical application in ~7 human studies of epithelial and stromal HSV keratitis with or without an adjuvant antiviral therapy. More importantly, PROKERA SLIM in conjunction with oral acyclovir has been shown to facilitate the ease of early intervention to accelerate restoration in herpetic keratitis in 2 case series of 5 eyes. However, a formal prospective study has not been performed.

ELIGIBILITY:
Inclusion Criteria:

1. The subject (male or female) is at least 18 years of age.
2. The subject is presenting with primary or recurrent herpetic dendritic epithelial keratitis based on investigator judgement
3. The subject is presenting with acute (within 30 days) herpetic dendritic epithelial keratitis
4. The subject is willing to comply with all study procedures and is able to consent.

Exclusion Criteria:

1. Clinical signs of a cause other than herpes simplex virus
2. Presence of corneal ulcer with or without microbial infection
3. Lid surface abnormalities or conjunctival scarring that affect lid function in either eye
4. Atopic disease
5. History of penetrating keratoplasty
6. Active stromal keratitis or iritis
7. Presence of systemic or ocular infection or inflammation that is not related to herpes simplex virus (such as Sarcoidosis, Cogan syndrome, atopy, Lyme disease, Syphilis, mumps, Epstein-Barr virus)
8. Ocular surface malignancy
9. History of recent ocular surgery/trauma, which could affect corneal sensitivity, e.g., corneal transplantation, LASIK
10. A medical or ocular condition, or a personal situation, which in the principal investigator's opinion, is not appropriate for participation in the trial
11. Current enrollment in another interventional drug or device study or participation in such a study within 30 days of anticipated entry into this study
12. Not capable of providing informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Time-dependent change in BCVA by 1 weeks | 1 week
  The BSCVA was recorded at 4 meters by a refractionist certified for the study using a protocol adapted from the Age-Related Eye Disease Study using Early Treatment Diabetic Retinopathy Study charts: chart R(2110), chart 1(2111), and chart 2(2112) (Precision Vision, Woodstock, IL).

SECONDARY OUTCOMES:
Proportion of patients with complete epithelialization by 1 week | 1 week
  Proportion of patients with complete epithelialization by 1 week, graded 0, SPK 1+, SPK 2+, SPK 3+ (SPK is Superficial Punctate Keratitis)
Time-dependent change in BCVA by 2 weeks | 2 weeks
  The BSCVA was recorded at 4 meters by a refractionist certified for the study using a protocol adapted from the Age-Related Eye Disease Study using Early Treatment Diabetic Retinopathy Study charts: chart R(2110), chart 1(2111), and chart 2(2112) (Precision Vision, Woodstock, IL).
Time-dependent change in BCVA by 2 months | 2 months
  The BSCVA was recorded at 4 meters by a refractionist certified for the study using a protocol adapted from the Age-Related Eye Disease Study using Early Treatment Diabetic Retinopathy Study charts: chart R(2110), chart 1(2111), and chart 2(2112) (Precision Vision, Woodstock, IL).
Proportion of patients with corneal opacity at 2 months | 2 months
  Proportion of patients with corneal opacity at 2 months, graded 0, 1+, 2+, 3+, and 4+.
Proportion of patients with recurrence by 2 months | 2 months
  Proportion of patients with recurrence by 2 months counted individually
Change in corneal sensitivity from baseline to 2 months | 2 months
  Change in corneal sensitivity from baseline to 2 months using Cochet-Bonnet esthesiometer, graded 0/4, 1/4, 2/4, 3/4, and 4/4.
Change in conjunctival inflammation at 1 week | 1 week
  Conjunctival inflammation graded by investigator as none (0), mild (1), moderate (2), and severe (3)
Change in conjunctival inflammation at 2 week | 2 week
  Conjunctival inflammation graded by investigator as none (0), mild (1), moderate (2), and severe (3)
Total number of extra patient visits, treatments, and procedures throughout study | 2-3 months
  Total number of extra patient visits, treatments, and procedures throughout study, counted individually by type

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stutzman, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute, Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Share EPD once available
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year